CLINICAL TRIAL: NCT00718068
Title: Assessing the Safety of a Continuous Potassium Chloride Infusion in Critical Care: A Randomised Controlled Trial
Brief Title: Safety of Continuous Potassium Chloride Infusion in Critical Care
Acronym: ASPIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Queen Elizabeth Hospital (Other)
Responsible Party: Dr Richard Chalwin, The Queen Elizabeth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007185
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2009-11

CONDITIONS: Hypokalemia; Arrhythmias, Cardiac
Keywords: Potassium chloride; Preparations, Pharmaceutical; Hypokalemia; Critical Care; Adult; Randomized Controlled Trial
MeSH Terms: conditions — Hypokalemia; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous (Experimental): This group will receive potassium chloride by continuous infusion on a sliding-scale system based on serum potassium level.
  Interventions: Drug: Sterile Potassium Chloride Concentrate
- Intermittent (Active Comparator): This arm will form the control group and receive potassium chloride by intermittent infusion as per conventional management
  Interventions: Drug: Sterile Potassium Chloride Concentrate

INTERVENTIONS:
Drug: Sterile Potassium Chloride Concentrate — Continuous infusion, 40mmol in 40ml, starting at 10ml/hr, rate altered according to serum potassium level checked 2 hourly
  Other Names: CAS no: 7447-40-7
  Arms: Continuous
Drug: Sterile Potassium Chloride Concentrate — By intermittent infusion, 20mmol diluted in 100ml 0.9% NaCl, administered over 60 mins, serum potassium level checked 2 hourly, and repeat doses administered as appropriate
  Other Names: CAS no: 7447-40-7
  Arms: Intermittent

SUMMARY:
Patients in critical care often require supplemental potassium chloride if levels in their blood are below acceptable level. Common practice is to administer a single dose of potassium chloride under controlled conditions via a drip, before checking if a further dose is required. The purpose of this study is to ensure that it is safe to administer potassium chloride continuously with the dose varied according to patient needs.

DETAILED DESCRIPTION:
The use of potassium supplementation is commonplace in the critical care environment. Patients often have abnormal serum potassium levels due to active disease processes. Conditions such as acute renal failure and metabolic acidosis precipitate hyperkalaemia, with ileus and insensible losses causing hypokalaemia. Both hypo- and hyperkalaemia can cause life-threatening arrythmias so it is prudent to rectify aberrant levels.

The standard treatment of hypokalaemia in intensive care units is by intravenous administration of potassium chloride. This can be given either as a dilute solution as maintenance intravenous fluid therapy, or as a concentrated solution by intermittent infusion. Alternatively potassium can be given as a concentrated solution by continuous infusion. All techniques require regular monitoring of the patient's serum potassium level with appropriate alterations to the administration regime.

From a theoretical standpoint it would make sense to give potassium by continuous infusion as this allow slow but steady correction of hypokalaemia. A continuous infusion should prevent rapid fluctuations in the serum level that could be caused by intermittent infusions, which may precipitate arrhythmia. However continuous infusions require vigilant monitoring to ensure that hyperkalaemia does not occur and must be given into a central vein to avoid the risk of phlebitis.

The use of intermittent infusions has been used safely in the critical care setting under physician guidance. A retrospective review reported the outcomes of the administration of 495 infusion sets to 190 individuals. While they identified 2 instances of post-infusion hyperkalaemia, neither was associated with any adverse sequelae. Analysis showed a no correlation between serum potassium increase post-infusion and serum creatinine, thus advocating the use of this therapy in patients with renal failure. In light of this valuable safety data, they proceeded with a prospective cohort study involving 40 patients on their Intensive Care Unit. Again the outcomes were favourable with a mean increase of 0.48mmol/L after administration of 20mmol in 100ml of saline over 1 hour. They reported no instances of hyperkalaemia, and data suggested a decreased instance of ectopic beats versus control patients.

The use of a variable dose regime dictated by serum potassium concentration has also been assessed. In a prospective cohort study 20, 30 or 40mmol was administered over 1 hour to 48 patients based on their initial measured potassium level. They only reported 2 instances of hyperkalaemia but neither patient experienced any complications. Usefully they found that patients with oliguric renal failure (creatinine 283 ± 127 micromol/L) had no greater mean increase in potassium level after infusion than patients with normal creatinine clearance.

Two other methods have been suggested. The first, assessed on a paediatric intensive care unit, administered potassium at a rate of 0.25mmol/kg/hr to patients with serum potassium < 3.5mmol/L and ECG abnormalities. The infusion was continued until the ECG abnormalities were corrected. Serum potassium wasn't measured until after completing the infusion, and although the mean increase was only 0.75mmol/L, this method did expose patients to a risk of unmonitored hyperkalaemia. The other involves use of a feedback system with a computer-algorithm driven protocol. This method was not developed into a full production model due to lack of cost-effectiveness.

We were unable to find any trials assessing the efficacy and safety of continuous potassium infusions in the critical care population, so felt it was time this was rectified. Critically ill patients are often hypokalaemic due to insensible losses, inadequate supplementation prior to admission, and use of diuretics and beta-agonists. At the same time they often have acute and/or chronic renal failure or may have a metabolic acidosis that will hamper normal potassium sequestration or excretion. Thus they are at risk of rapidly developing life-threatening hyperkalaemia if supplementation is not carefully titrated against serial monitoring. Continuous infusions administered with due vigilance should allow for correction of hypokalaemia in a safe and precise manner.

Our department used to supplement potassium by intermittent infusion, but after internal discussion we have successfully implemented a continuous infusion protocol. We propose that continuous infusions administered by accredited nurses under physician direction can safely deliver potassium and correct abnormal levels.

ELIGIBILITY:
Inclusion Criteria:

* Any inpatient on the investigating unit with a serum potassium level of less than 3.8mmol/L
* arterial line for blood sampling and central venous access for infusion administration in situ
* continuous 12-lead ECG monitoring

Exclusion Criteria:

* Patients with a serum potassium ≥ 3.8mmol/L
* Renal dysfunction with serum creatinine 50% greater than the upper end of the normal reference range (i.e.: > 180micromol/L) or urine output less than 0.5ml/kg/hr for 6 consecutive hours, or the requirement for dialysis
* Burns
* Hypomagnesaemia (≤ 0.7mmol/L), however patients may be enrolled after the hypomagnesaemia is corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-10; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Adherence to a potassium level 4.0 - 4.5mmol/L | 7 days

SECONDARY OUTCOMES:
Total quantity of potassium administered | 7 days
Incidence of potassium level < 3.0mmol/L and > 5.5mmol/L | 7 days
Incidence of arrhythmia | 7 days
Number of arterial blood gases taken | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chalwin, FCICM, Principal Investigator — The Queen Elizabeth Hospital
Locations (1):
- The Queen Elizabeth Hospital, Woodville South, South Australia, Australia